CLINICAL TRIAL: NCT03056287
Title: Treating Depression and Enhancing Locomotor Recovery Post-stroke
Brief Title: Exercise and Brain Stimulation for Post-stroke Depression
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of South Carolina (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Treatment
Other Study IDs: COBRE: EXD
Record Dates: First submitted 2017-02-08; First posted 2017-02-17 (Actual); Results first posted 2025-05-14 (Actual); Last update posted 2025-05-14 (Actual); Status verified 2025-05

CONDITIONS: Stroke
MeSH Terms: conditions — Stroke | interventions — Exercise; Transcranial Magnetic Stimulation

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Aerobic Exercise (Experimental): Treadmill aerobic exercise
  Interventions: Behavioral: Aerobic exercise
- rTMS (Experimental): repetitive transcranial magnetic stimulation
  Interventions: Other: Repetitive transcranial magnetic stimulation
- AET+rTMS (Experimental): Combined aerobic exercise and rTMS
  Interventions: Behavioral: Aerobic exercise; Other: Repetitive transcranial magnetic stimulation
- Sham (Sham Comparator): Sham rTMS
  Interventions: Other: Repetitive transcranial magnetic stimulation

INTERVENTIONS:
Behavioral: Aerobic exercise — treadmill aerobic exercise; 3 sessions per week, 40 minutes per session
  Arms: AET+rTMS; Aerobic Exercise
Other: Repetitive transcranial magnetic stimulation — Repeated non-invasive brain stimulation to the left dorsolateral prefrontal cortex.
  Other Names: rTMS
  Arms: AET+rTMS; Sham; rTMS

SUMMARY:
This project will assess the effects of aerobic exercise training (AET), repetitive transcranial magnetic stimulation (rTMS) or their combination on depressive severity as well as locomotor function in persons with post-stroke depression (PSD). Both AET and rTMS are established stand-alone treatments for non-stroke related depression, though neither has been adequately studied post-stroke. Furthermore, substantive research indicates that AET improves post-stroke locomotor function, thus offering a novel approach for treating PSD as well as an established vehicle to study the effects of PSD on response to rehabilitation.

The purpose of this project is to determine the impact of AET, rTMS and their combination (AET+rTMS) treatments on post-stroke depressive symptoms and locomotor function so as to guide the development of a future clinical trial. A total of 40 depressed post-stroke subjects will be randomly assigned to one of four groups 1) AET; 2) rTMS; 3) combined AET and rTMS (AET+rTMS) or 4) control (sham rTMS) group (n=10 per condition; equally distributed with mild and moderate MDD). Further, an additional 10 non-depressed post-stroke subjects will complete 8 weeks of AET so as to allow us to determine the effects of PSD on response to training (Aim 2). Training (AET, rTMS and AET+rTMS) will take place over an 8-week period, three times per week on non-consecutive days. Measures of depression (HRSD17) as well as self-selected walking speed (SSWS) will be performed prior to the initial treatment session of each week as well as 8 weeks following cessation of treatment. Additional measures of locomotor function (walking endurance and amount of daily community stepping) will be assessed prior to training (pre), following 4 weeks of training (mid), upon completion of 8 weeks of training (post) as well as 8 weeks following cessation of training (follow-up), allowing determination of the efficacy (and persistence) of training on these outcomes.

ELIGIBILITY:
Inclusion Criteria:

1. age 50-70
2. stroke within the past 6 to 60 months,
3. major depressive disorder (PHQ-9 > 10) and diagnosed using the Structured Clinical Interview for Depression (SCID) according to the Diagnostic and Statistical Manual of Mental Disorders, Fourth Edition (DSM-IV),
4. residual paresis in the lower extremity (Fugl-Meyer LE motor score <34),
5. ability to walk without assistance and without an AFO on the treadmill ≥ 30 seconds at speeds ranging from 0.2-0.8 m/s,
6. no antidepressant medications or clinically able to discontinue medications,
7. HRSD question #9 regarding suicide <2,
8. provision of informed consent. In addition, all subjects who meet criteria for the training portion must complete an exercise tolerance test and be cleared for participation by the study cardiologist.

Exclusion Criteria:

1. Unable to ambulate at least 150 feet prior to stroke, or experienced intermittent claudication while walking;
2. history of congestive heart failure, unstable cardiac arrhythmias, hypertrophic cardiomyopathy, severe aortic stenosis, angina or dyspnea at rest or during ADL's;
3. History of oxygen dependence;
4. Preexisting neurological disorders, dementia or previous stroke;
5. History of major head trauma;
6. Legal blindness or severe visual impairment;
7. history of psychosis or other Axis I disorder that is primary;
8. Life expectancy <1 yr.;
9. Severe arthritis or other problems that limit passive range of motion;
10. History of DVT or pulmonary embolism within 6 months;
11. Uncontrolled diabetes with recent weight loss, diabetic coma, or frequent insulin reactions;
12. Severe hypertension with systolic >200 mmHg and diastolic >110 mmHg at rest;
13. attempt of suicide in the last 2 years or at suicidal risk assessed by SCID interview;
14. Previous or current enrollment in a clinical trial to enhance motor recovery;
15. currently exercising ≥ 2 times per week (≥20 minutes);
16. Presence of non-MR compatible implants, pregnancy or severe claustrophobia.

Ages: 50 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 23 (Actual)
Dates: Start 2016-01-01 (Actual); Primary Completion 2019-12-31 (Actual); Study Completion 2019-12-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Chris M Gregory, PhD, Principal Investigator — Medical University of South Carolina
Locations (1):
- Medical University of South Carolina, Charleston, South Carolina, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Aerobic Exercise | rTMS | AET+rTMS | Sham
Started | 4 | 6 | 6 | 7
Completed | 4 | 5 | 5 | 6
Not Completed | 0 | 1 | 1 | 1
Not completed — Withdrawal by Subject | 0 | 1 | 0 | 0
Not completed — move out of area | 0 | 0 | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Aerobic Exercise | rTMS | AET+rTMS | Sham | Total
Number analyzed (Participants) | 4 | 6 | 6 | 7 | 23
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 4 | 3 | 4 | 6 | 17
  >=65 years | 0 | 3 | 2 | 1 | 6
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 4 | 3 | 4 | 14
  Male | 1 | 2 | 3 | 3 | 9
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 3 | 1 | 3 | 3 | 10
  White | 1 | 5 | 3 | 4 | 13
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 4 | 6 | 6 | 7 | 23

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline to Post Training in Hamilton Rating Scale for Depression
Description: The Hamilton Rating Scale for Depression is a clinician-administered depression assessment scale containing 17 items pertaining to symptoms of depression experienced over the past week. A total score of 0-7 is generally accepted to be within the normal range (or in clinical remission), while a total score of 20 or higher indicates at least moderate severity depression. Score range 0-58. Higher total scores indicate higher levels of depression, while a score of 0 would indicate no depressive symptoms.
Time Frame: assessed at baseline and weekly throughout the 8 week intervention. Change from baseline to week 8 reported as primary outcome
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Aerobic Exercise | rTMS | AET+rTMS | Sham
Number analyzed (Participants) | 4 | 6 | 6 | 7
units on a scale | -2.75 (4.5) | -7.5 (5.46) | -7.83 (4.49) | -2.29 (2.63)

2. Secondary Outcome: Change From Baseline to Week 8 in Self-selected Walking Speed
Time Frame: assessed at baseline as well as weekly throughout the 8 week intervention. Change from baseline to week 8 reported as outcome
Measure: Mean (Standard Deviation); unit: centimeters per second
Arm/Group | Aerobic Exercise | rTMS | AET+rTMS | Sham
Number analyzed (Participants) | 4 | 6 | 6 | 7
centimeters per second | 8.2 (9.52) | 7.7 (15.43) | 30.65 (20.24) | 2.19 (15.04)

ADVERSE EVENTS:
Time Frame: Throughout the 8 week intervention as well as during an 8 week follow-up period. Collected over a total of weeks
Arm/Group | Aerobic Exercise | rTMS | AET+rTMS | Sham
All-Cause Mortality (participants affected / at risk) | 0/4 | 0/6 | 0/6 | 0/7
Serious Adverse Events (participants affected / at risk) | 0/4 | 0/6 | 0/6 | 0/7
Other Adverse Events (participants affected / at risk) | 1/4 | 0/6 | 1/6 | 0/7
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Aerobic Exercise (N=4) | rTMS (N=6) | AET+rTMS (N=6) | Sham (N=7)
fall (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) — minor fall

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-02-28): https://cdn.clinicaltrials.gov/large-docs/87/NCT03056287/Prot_SAP_000.pdf